CLINICAL TRIAL: NCT07155278
Title: Efficacy and Safety of a Particulated Human Acellular Dermal Matrix Skin Booster: A Randomized, Split-Face, Double-blinded, Prospective Clinical Trial
Brief Title: Efficacy & Safety of hADM Skin Booster
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Korea International Cooperation Agency (KOICA) (Unknown)
Responsible Party: Principal Investigator, Ngoc Ha Nguyen, Dr., Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-2024-0042
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Rhytides; Skin Texture Irregularities; Photoaged Facial Skin; Skin Lifting and Tightening
Keywords: Acellular dermal matrix; Dermal filler; Skin booster; Hyaluronic acid; Skin rejuvenation

STUDY DESIGN:
Intervention Model Description: Each right or left side of the eligible participants' faces was randomly assigned one of the two treatment arms. The test side of each participant's face received a combination of Elravie Re2O (containing phADM) and Elravie Balance (Hyaluronic acid), while the control side received only Elravie Balance.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm A (Experimental): One randomly assigned half of each participant's face received a combination of Elravie Re2O (phADM) and Elravie Balance (hyaluronic acid).
  Interventions: Drug: Elravie Re2O; Drug: Elravie Balance
- Treatment arm B (Active Comparator): The remaining half of each participant's face received Elravie Balance (hyaluronic acid) only.
  Interventions: Drug: Elravie Balance

INTERVENTIONS:
Drug: Elravie Re2O — Elravie Re2O is a particulated human Acellular Dermal Matrix (phADM), with each 5 mL syringe containing 150 mg of phADM. This product is classified as a human tissue product and received its approval via a tissue bank establishment permit from the Ministry of Food and Drug Safety.
  Arms: Treatment arm A
Drug: Elravie Balance — Elravie Balance is a gel-type hyaluronic acid (HA) skin booster. It contains HA at a concentration of 20mg/ml in a 2.5 cc syringe with a volume of 1.5 mL.

SUMMARY:
The goal of this randomized, split-face, double-blinded clinical trial is to evaluate the efficacy and safety of Elravie Re2O (particulated human Acellular Dermal Matrix, phADM) as a skin booster compared with hyaluronic acid (HA) skin booster alone in adults with skin roughness.

The main questions it aims to answer are:

1. Does phADM combined with HA improve objective skin measurements and subjective skin assessments more effectively than HA alone?
2. Is phADM + HA treatment safe and well tolerated?

Researchers will compare one half of participant's face treated with phADM + HA versus the opposite cheek treated with HA alone to see if phADM provides superior skin improvement.

Participants will:

1. Be randomly assigned to receive three intradermal injections at one-month intervals, with phADM + HA on one cheek and HA alone on the other.
2. Undergo follow-up visits over 20 weeks for evaluation of ACSS score, instrumental skin quality measurements (e.g., skin density, volume, wrinkles), and satisfaction (GAIS).
3. Be monitored for local adverse events and changes in vital signs to assess safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 30 to 65 years old
* Those with an Allergan Cheek Smoothness Scale (ACSS) score of 2-3 during screening

Exclusion Criteria:

* Those who have received dermal fillers, botulinum toxin injections, mesotherapy, or other cosmetic procedures (e.g., laser) on the face within 12 months of screening or plan to receive such treatments during the trial period.
* Those who received facial wrinkle correction treatment within 6 months of screening
* Those with inflammatory diseases in the facial area
* Those with infectious diseases, skin grafts, keloids, or hypertrophic scars on the face.
* Those with autoimmune diseases
* Those who have experienced anaphylaxis or severe complex allergies for any reason
* Those who were prescribed anticoagulant therapy within 2 weeks of the screening date
* Those with a history of serious cardiopulmonary disease
* Breastfeeding
* Those who have started using or taking external or oral agents for wrinkle improvement within 30 days of screening

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Nasolabial fold depth | Baseline and 1, 4, 8, 12, 16, and 20 weeks post-treatment
  Nasolabial fold depth was measured using the Antera 3D CS (Miravex, Dublin, Ireland), which quantifies wrinkle depth in millimeters (mm)
Under-eye wrinkles | Baseline and 1, 4, 8, 12, 16, and 20 weeks post-treatment
  The Eve V (EVELAB INSIGHT, Singapore) was used to measure under-eye wrinkles in pixels.
Skin volume | Baseline and 1, 4, 8, 12, 16, and 20 weeks post-treatment
  Skin volume was measured in cubic millimeters (mm3) with the 3D LifeViz micro (QuantifiCare, Biot, France)
Skin density | Baseline and 1, 4, 8, 12, 16, and 20 weeks post-treatment
  Skin density was evaluated in percentage (%) using the Skin Scanner (tpm, Luneburg, Germany)
Pore area | Baseline and 1, 4, 8, 12, 16, and 20 weeks post-treatment
  Pore area was measured using the Antera 3D CS (Miravex, Dublin, Ireland), which quantifies pore area in millimeters squared (mm2).
Eye and cheek area lifting | Baseline and 1, 4, 8, 12, 16, and 20 weeks post-treatment
  Eye and cheek area lifting was assessed with the Morpheus3D (Morpheus, Gyeonggi, Republic of Korea),which measures the increase in curve length in millimeters to determine the degree of lifting.

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale | Baseline and 1, 4, 8, 12, 16, and 20 weeks post-treatment
Allergan Cheek Smoothness Scale | Baseline and 1, 4, 8, 12, 16, and 20 weeks post-treatment

OTHER OUTCOMES:
Adverse event assessment | From baseline to 20 weeks post-treatment
  The safety of the test products was assessed throughout the study period. During each visit, participants were monitored for any adverse reactions, and the use of any concomitant medications that could potentially affect the study was checked. All confirmed and reported adverse reactions from all subjects were compiled to determine the incidence rate, which was then used as data for the overall safety evaluation of the product.

CONTACTS AND LOCATIONS:
Overall Officials: Ju Hee Lee, M.D., Ph.D., Principal Investigator — Department of Dermatology & Cutaneous Biology Research Institute, Yonsei University College of Medicine, Seoul, Republic of Korea
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional policies that restrict data sharing beyond the research team. Data were collected under a protocol that did not include participant consent for public or external data sharing.